CLINICAL TRIAL: NCT04322032
Title: A Randomized, Open-label, Single Dose, Crossover Study to Evaluate the Pharmacokinetic Profiles and Safety of CKD-389 in Healthy Volunteers Under Fasting Conditions
Brief Title: Clinical Study to Evaluate the Pharmacokinetic Profiles and Safety of CKD-389
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A102_02BE2003
Record Dates: First submitted 2020-03-24; First posted 2020-03-26 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Drug Evaluation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): 1. Period 1: Reference drug
  2. Period 2: Test drug
  Interventions: Drug: Reference drug; Drug: Test drug
- Group 2 (Experimental): 1. Period 1: Test drug
  2. Period 2: Reference drug
  Interventions: Drug: Reference drug; Drug: Test drug

INTERVENTIONS:
Drug: Reference drug — D759 Tab. 1 Tab. and D308 Tab. 1 Tab.(Total 2 Tab.), Single oral administration under fasting condition.
  Other Names: D759 and D308
Drug: Test drug — CKD-389 Tab. 1 Tab.(Total 1 Tab.), Single oral administration under fasting condition.
  Other Names: CKD-389

SUMMARY:
This study is a randomized, open-label, fasted, single dose, crossover study to evaluate the pharmacokinetic profiles and safety of CKD-389 in healthy volunteers.

DETAILED DESCRIPTION:
To healthy subjects of thirty-four (34), following treatments are administered dosing in each period and wash-out period is a minimum of 7 days. Reference drug(D759 and D308), Test drug(CKD-389) Pharmacokinetic blood samples are collected up to 48 hrs. The pharmacokinetic characteristics and safety are assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults over the age of 19 years and under the age of 65 years at the time of screening
2. Subject who had 17.5kg/m² ≤ Body Mass Index (BMI) < 30.5kg/m² and a total body weight of males ≥ 55 kg and females ≥ 45 kg

   # BMI=Weight(kg) / Height(m)²
3. Subject without congenital/chronic diseases and without abnormal symptoms or diagnosis based on a medical examination within the last 3 years
4. Subject who were deemed to be appropriate as study subjects in accordance with the screening results (laboratory tests, vital signs, ECG etc.)
5. Subject who signed an informed consent form approved by the Institutional Review Board(IRB) of Chonbuk National University Hospital and decided to participate in the study after being fully informed of the study prior to participation, including the objective, content and characteristics of the investigational drug
6. Subject who consents to the use of reliable contraception during the clinical trial and not to donate his sperm during the study period and until 1 month after the last administration of investigational product
7. Subject with the ability and willingness to participate during the study period

Exclusion Criteria:

1. Subjects with a medical evidence or a history (excluding a dental history of periodontal surgery, impacted wisdom teeth removal, etc.) of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, urinary, cardiovascular, hepatic, psychiatric, neurologic or immune disease
2. Subjects with a medical history of gastrointestinal disease (e.g., gullet disease such as esophageal achalasia and esophagostenosis and Crohn's disease) or operations (excluding simple appendectomy, herniotomy or tooth extraction) that may affect drug absorption
3. Subjects with the following laboratory test result:

   ☞ ALT or AST > 2x the upper limit of the normal range
4. History of regular alcohol consumption exceeding 210 g/week within 6 months prior to screening (1 drink (250 mL) of beer (5%) = 10 g; 1 drink (50 mL) of hard liquor (20%) = 8 g; 1 drink (125 mL) of wine (12%) = 12 g)
5. Subjects who smoked more than 20 cigarettes per day within 6 months prior to screening
6. Subjects who had been administered investigational product(s) from other clinical study or bioequivalence study within 6 months prior to the first dose of this study
7. Following vital signs at screening

   ☞ Sitting systolic blood pressure ≥160 mmHg or <90 mmHg and/or a sitting diastolic blood pressure ≥100 mmHg or <50 mmHg at screening
8. Subjects with a medical history of significant alcohol or drug abuse within one year prior to the screening
9. Subjects who had taken any drug(s) known as a strong inducer(s) or inhibitor(s) of drug-metabolizing enzymes within 30 days prior to the first dose of investigational product(s)
10. Subjects who had taken prescription or nonprescription drugs within 10 days prior to the first dose of investigational product(s)
11. Subjects who donated whole blood within 2 months or blood components within 1 month prior to the first dose of the investigational product(s)
12. Subjects with a severe acute/chronic physical and mental conditions that can increase risk or interfere with the interpretation of the results of test
13. Subjects who had Type 1 diabetes or diabetic ketoacidosis
14. Subjects with known hypersensitivity to the drug or the drug ingredient, such as anaphylactic reactions or angioedema
15. Subject had renal impairment(eGFR < 60 mL/min/1.73 m²)
16. Subject had genetic dysfunctions like galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption
17. Subject who is a pregnant or nursing woman
18. Subject had heart failure(NYHA class IV)
19. Subjects who were deemed inappropriate to participate in the study by the investigator

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2020-04-06 (Estimated); Primary Completion 2020-05-12 (Estimated); Study Completion 2020-05-18 (Estimated)

PRIMARY OUTCOMES:
AUCt(Area Under Curve last) | Each period: Pre-dose (0 hour), post-dose 0.17, 0.33, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48 h
  Area under the plasma concentration time curve of CKD-389/D759&D308, from time zero up to the last measurable concentration.
Cmax | Each period: Pre-dose (0 hour), post-dose 0.17, 0.33, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48 h
  The maximum concentration observed of CKD-389/D759&D308 over blood sampling time.

CONTACTS AND LOCATIONS:
Overall Officials: Min-gul Kim, Principal Investigator — Chonbuk National University Hospital
Locations (1):
- Chonbuk National University Hospital, Jeonju, South Korea

IPD SHARING:
Plan to Share IPD: No